CLINICAL TRIAL: NCT05028868
Title: Clinical Research of Intravenous Thrombolysis for Ischemic Stroke in Northeast of China
Acronym: CRISTINA
Status: Recruiting | Type: Observational
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Associate dean, Director of Cerebrovascular Disease Center, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Other Study IDs: CRISTINA
Record Dates: First submitted 2017-03-07; First posted 2021-08-31 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Ischemic Stroke; Thrombosis
Keywords: ischemic stroke; thrombolysis
MeSH Terms: conditions — Ischemic Stroke; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (5):
- Large artery atherosclerosis(LAA)
- Cardiogenic stroke(CS)
- Penetrating artery disease(PAD)
- Other etiology(OE)
- undetermined etiology(UE)

SUMMARY:
This research is based on clinic treatment of intravenous thrombolysis for patients with acute ischemic stroke.By building up a database of these patients, the investigators aim to find some significance between groups by analyzing population information, clinical status and such for better evaluation and optimal treatment decision.

DETAILED DESCRIPTION:
With the highest incidence rate,the population in northeast of China is severely tormented by stroke, especially ischemic stroke. The investigators lunch this project by building up a database of detailed information of patients that fits the criteria of intravenous thrombolysis therapy.Including biochemical markers,imaging and follow-up,investigators intend to analysis these data,find factors that contributes to better prognosis,so as to push forward the prevention and control work.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of ischemic stroke causing measurable neurological deficit
2. Onset of symptoms <4.5 h before treatment begins
3. Age ≥18 y

Exclusion Criteria:

1. Significant head trauma or prior stroke in the previous 3 mo
2. Symptoms suggest SAH
3. Arterial puncture at noncompressible site in previous 7 d
4. History of previous intracranial hemorrhage
5. Intracranial neoplasm, AVM, or aneurysm
6. Recent intracranial or intraspinal surgery
7. Elevated blood pressure (systolic >185 mm Hg or diastolic >110 mm Hg)
8. Active internal bleeding
9. Acute bleeding diathesis, including but not limited to
10. Platelet count <100 000/mm3
11. Heparin received within 48 h resulting in abnormally elevated aPTT above the upper limit of normal
12. Current use of anticoagulant with INR >1.7 or PT >15 s
13. Current use of direct thrombin inhibitors or direct factor Xa inhibitors with elevated sensitive laboratory tests (eg, aPTT, INR, platelet count, ECT, TT, or appropriate factor Xa activity assays)
14. Blood glucose concentration <50 mg/dL (2.7 mmol/L)
15. CT demonstrates multilobar infarction (hypodensity >1/3 cerebral hemisphere)
16. Relative exclusion criteria
17. Recent experience suggests that under some circumstances, with careful consideration and weighting of risk to benefit, patients may receive fibrinolytic therapy despite ≥1 relative contraindications. Consider risk to benefit of intravenous rtPA administration carefully if any of these relative contraindications is present
18. Only minor or rapidly improving stroke symptoms (clearing spontaneously)
19. Pregnancy
20. Seizure at onset with postictal residual neurological impairments
21. Major surgery or serious trauma within previous 14 d
22. Recent gastrointestinal or urinary tract hemorrhage (within previous 21 d)
23. Recent acute myocardial infarction (within previous 3 mo)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute ischemic stroke within 4.5h from symptoms onset who received IV rt-PA.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-06-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2026-01-28 (Estimated)

PRIMARY OUTCOMES:
mRS score in 90 days | 90 days
  Using mRS score to evaluate the effective of thrombolysis among different groups.
Stroke recurrence within 90 days | 90 days
  Newly onset stroke that the time interval was less than 90 days from the original stroke event was considered as stroke recurrence. Ischemic stroke was defined as acute focal brain or retinal infarction.

SECONDARY OUTCOMES:
Cardiovascular death in 1 year | 1 year
  Death direct from ischemic stroke, hemorrhagic stroke, sudden cardiac death, acute myocardial infarction, heart failure, and other cardiovascular death including cardiac arrhythmia that unrelated to sudden cardiac death, pulmonary embolism, cardiovascular intervention (unrelated to acute MI), ruptured aortic aneurysm, or peripheral arterial disease).
Post-stroke disability in 1 year | 1 year
  modified Rankin Scale(mRS)≥3

CONTACTS AND LOCATIONS:
Overall Officials: Yi Yang, MD，PhD, Study Chair — The First Hospital of Jilin University
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang HM, Shen ZD, Qu Y, Zhang P, Abuduxukuer R, Wang LJ, Li Y, Chen YM, Liu AR, Liu XD, Zhao LL, Yang CY, Yao J, Wang AY, Jiang YF, Wang JC, Dong CP, Liu FF, Li L, Qi YB, Wang CF, Li H, Zhang LY, Ma WJ, Guo ZN, Yang Y. External validation of N2H3 nomogram to predict outcomes in patients with acute ischemic stroke treated by intravenous thrombolysis. Brain Circ. 2025 Mar 4;11(3):212-218. doi: 10.4103/bc.bc_81_24. eCollection 2025 Jul-Sep. PMID 40842451